CLINICAL TRIAL: NCT01934127
Title: An Observer-blind Study to Evaluate the Safety and Immunogenicity of GSK Biologicals' Influenza Vaccine(s) GSK2789869A and GSK2789868A Administered in Adults 21 to 64 Years of Age
Brief Title: Immunogenicity and Safety Study of Different Formulations of GlaxoSmithKline (GSK) Biologicals H7N1 Influenza Vaccine Administered to Adults 21 to 64 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 115415
Record Dates: First submitted 2013-08-01; First posted 2013-09-04 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Influenza
Keywords: Immunogenicity; H7N1; Influenza; Safety; AS03 adjuvant; Adults
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- Formulation 1 Group (Experimental): Subjects in this group will receive two doses of GSK2789869A H7N1 vaccine formulation 1 at a 21 day interval
  Interventions: Biological: Investigational H7N1 vaccine GSK2789869A
- Formulation 2 Group (Experimental): Subjects in this group will receive two doses of GSK2789869A H7N1 vaccine formulation 2 at a 21 day interval
  Interventions: Biological: Investigational H7N1 vaccine GSK2789869A
- Formulation 3 Group (Experimental): Subjects in this group will receive two doses of GSK2789869A H7N1 vaccine formulation 3 at a 21 day interval
  Interventions: Biological: Investigational H7N1 vaccine GSK2789869A
- Formulation 4 Group (Experimental): Subjects in this group will receive two doses of GSK2789869A H7N1 vaccine formulation 4 at a 21 day interval
  Interventions: Biological: Investigational H7N1 vaccine GSK2789869A
- Formulation 5 Group (Experimental): Subjects in this group will receive two doses of GSK2789868A H7N1 vaccine formulation 5 at a 21 day interval
  Interventions: Biological: Investigational H7N1 vaccine GSK2789868A
- Placebo Group (Placebo Comparator): Subjects in this group will receive two doses of placebo at a 21 day interval
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Investigational H7N1 vaccine GSK2789869A — One dose of GSK2789869A H7N1 vaccine administered intramuscularly at the deltoid region of the non-dominant arm at Day 0 while second dose of GSK2789869A H7N1 vaccine administered intramuscularly at the deltoid region of the dominant arm at Day 21
  Arms: Formulation 1 Group; Formulation 2 Group; Formulation 3 Group; Formulation 4 Group
Biological: Investigational H7N1 vaccine GSK2789868A — One dose of GSK2789868A H7N1 vaccine administered intramuscularly at the deltoid region of the non-dominant arm at Day 0 while the second dose of GSK2789868A H7N1 vaccine administered intramuscularly at the deltoid region of the dominant arm at Day 21
  Arms: Formulation 5 Group
Biological: Placebo — One dose of placebo administered intramuscularly at the deltoid region of the non-dominant arm at Day 0 while the second dose of placebo administered intramuscularly at the deltoid region of the dominant arm at Day 21
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of different formulations of GSK Biologicals H7N1 influenza vaccine in subjects 21 to 64 years of age. The study will evaluate safety related events and antibody immune responses to different formulations of study vaccine and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults who are 21 to 64 years of age (inclusive) at the time of first study vaccination.
* Written informed consent obtained from the subject.
* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Healthy subjects as established by medical history and physical examination.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or other multiple-user device.
* For subjects who undergo a screening visit, results of all safety laboratory tests obtained at the screening visit must be within reference ranges. Results of any repeat testing cannot be used to qualify a subject for enrollment.
* Female subjects of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if they

  * have practiced adequate contraception for 30 days prior to vaccination, and
  * have a negative pregnancy test on the day of vaccination, and
  * agree to continue to practice adequate contraception until 2 months after the last dose administered.

Exclusion Criteria:

* Presence or evidence of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence or evidence of substance abuse.
* Diagnosed with cancer, or treatment for cancer within three years.

  1. Persons with a history of cancer who are disease-free without treatment for three years or more are eligible.
  2. Persons with a history of histologically-confirmed basal cell carcinoma of the skin successfully treated with local excision only are excepted and are eligible, but other histologic types of skin cancer are exclusionary.
  3. Women who are disease-free three years or more after treatment for breast cancer and receiving long-term prophylaxis are eligible.
* Diagnosed with excessive daytime sleepiness (unintended sleep episodes during the day present almost daily for at least one month), or narcolepsy.
* History of narcolepsy in subject's parent, sibling or child
* Presence of a temperature ≥ 38.0ºC (≥100.4ºF), or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.

NOTE: The subject may be vaccinated at a later date, provided symptoms have resolved, and all other eligibility criteria continue to be satisfied.

* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Receipt of systemic glucocorticoids within 30 days prior to the first dose of study vaccine/placebo, or any other cytotoxic, immunosuppressive or immune-modifying drugs within 6 months of first study vaccine/ placebo dose. Topical, intra-articularly injected, or inhaled glucocorticoids, topical calcineurin inhibitors or imiquimod are allowed.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination are eligible. Persons receiving prophylactic antiplatelet medications, e.g., low-dose aspirin, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or Guillain Barré Syndrome within 42 days of receipt of prior seasonal or pandemic influenza vaccine.
* Administration of an inactive vaccine within 14 days or of a live attenuated vaccine within 30 days before the first dose of study vaccine/placebo.
* Planned administration of any vaccine other than the study vaccine/placebo before blood sampling at the Day 42 visit.
* Previous administration of any H7 vaccine or physician-confirmed H7 disease.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine/placebo, or planned use during the study period.
* Receipt of any immunoglobulins and/or any blood products within 90 days before the first dose of study vaccine/placebo, or planned administration of any of these products during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines or component used in the manufacturing process of the study vaccine including a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin (β-hCG) test result before the first dose of study vaccine/placebo.
* Lactating or nursing women.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 427 (Actual)
Dates: Start 2013-08-26 (Actual); Primary Completion 2013-11-01 (Actual); Study Completion 2014-10-20 (Actual)

PRIMARY OUTCOMES:
Humoral immune response in terms of vaccine-homologous hemagglutination inhibition (HI) antibody titers for each adjuvanted H7N1 vaccine group | At Day 42
  The following aggregate variables will be calculated: Seroconversion rates (SCR); Seroprotection rates (SPR); Mean Geometric Increase (MGI);
Occurrence of each solicited local symptom | During a 7-day follow-up period (i.e., day of vaccination and 6 subsequent days) after each vaccination
Occurrence of each solicited general symptom | During a 7-day follow-up period (i.e., day of vaccination and 6 subsequent days) after each vaccination
Occurrence of clinical safety laboratory abnormalities reported for samples | From Day 0 - 42 after each vaccination (i.e Days 0, 7 , 21, 28, 42)
Occurrence of unsolicited adverse events | 21 days after each dose
Occurrence of Medically Attended Adverse Events (MAEs), potential Immune Mediated Diseases (pIMDs) and Serious Adverse Events (SAEs) | From Day 0 until the Day 42 visit

SECONDARY OUTCOMES:
Humoral immune response in terms of Geometric mean reciprocal serum HI antibody titers (GMTs ratios) | At Day 42
  GMT ratios will be calculated for each adjuvanted (GSK2789869A) vaccine group which successfully meets Center for Biologics Evaluation and Research (CBER) and Committee for Medicinal Products for Human Use (CHMP) criteria, and for the unadjuvanted (GSK2789868A) plain antigen vaccine group
Humoral immune response in terms of vaccine-homologous HI antibody titers for the unadjuvanted (GSK2789868A) plain antigen vaccine group | At Day 42
  The following aggregate variables will be calculated : • SCR; • SPR; • MGI;
Vaccine-homologous (H7N1) HI antibody titers | • GMTs and Seropositivity rates at Days 0, 21, 42 and Months 6 and 12. • SCR and MGI at Day 21, 42 (Placebo group only) and Months 6 and 12. • SPR at Days 0, 21, 42 (Placebo group only) and Months 6 and 12.
  The following aggregate variables will be calculated for each study group: • GMTs; • Seropositivity rates; • SCR; • SPR; • MGI;
Vaccine-homologous (H7N1) HI antibody titers by age stratum | • GMTs, Seropositivity rates and SPR at Days 0, 21, 42 and Months 6 and 12. • SCR and MGI at Day 21, 42 and Months 6 and 12.
  The following aggregate variables will be calculated for each study group by age stratum (21-40 years; 41-64 years): • GMTs; • Seropositivity rates; • SCR; • SPR; • MGI;
Vaccine-heterologous (H7N9) HI antibody titers | • GMTs and Seropositivity rates and SPR at Days 0, 21, 42 and Months 6 and 12. • SCR and MGI at Day 21, 42 and Months 6 and 12.
Vaccine homologous (H7N1) and heterologous (H7N9) neutralizing (MN) antibody titers | • GMTs and Seropositivity rates at Days 0, 21, 42 and Month 6. • VRR at Days 21, 42 and Month 6.
Occurrence of MAEs, pIMDs and SAEs | After the Day 42 visit until the Month 12 visit
Humoral immune response in terms of SCR difference | At Day 42
  SCR difference will be calculated for each adjuvanted (GSK2789869A) vaccine group which successfully meets CBER and CHMP criteria, and for the unadjuvanted (GSK2789868A) plain antigen vaccine group

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- United States (6):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Austin, Texas
- Canada (3):
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Madan A, Ferguson M, Sheldon E, Segall N, Chu L, Toma A, Rheault P, Friel D, Soni J, Li P, Innis BL, Schuind A. Immunogenicity and safety of an AS03-adjuvanted H7N1 vaccine in healthy adults: A phase I/II, observer-blind, randomized, controlled trial. Vaccine. 2017 Mar 7;35(10):1431-1439. doi: 10.1016/j.vaccine.2017.01.054. Epub 2017 Feb 7. PMID 28187952
- See also: Results for study 115415 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/115415?search=study&#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 115415 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115415 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115415 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115415 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115415 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115415 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register